CLINICAL TRIAL: NCT01417832
Title: Radiographic Progression of Sealed and Infiltrated Caries Lesions in Vivo
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad El Bosque, Bogotá (Other)
Collaborators: DMG, Germany (Unknown)
Responsible Party: Universidad El Bosque, Bogotá, Stefania Martignon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOC_20080328131018
Record Dates: First submitted 2011-07-05; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Dental Caries
Keywords: Dental caries; Proximal surfaces; Preventive therapy; Dental radiography; Treatment efficacy; Young adults
MeSH Terms: conditions — Dental Caries | interventions — Adhesives; CMW cement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment with Infiltrant/Adhesive (Experimental): In this split-mouth design study, one of the three randomly selected approximal lesions will be treated with an infiltrant resin, one will be treated with an adhesive resin.
  Interventions: Drug: Resin infiltration / adhesive
- Placebo, placebo treatment (Placebo Comparator): In this split-mouth design study, one of the three randomly selected approximal lesions will be treated with a placebo treatment: At baseline one caries lesion was cleaned with a microbrush for 30 seconds and the procedure was repeated after two minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resin infiltration / adhesive — Treatment at baseline of one caries lesion with a resin infiltration conducted under rubber-dam isolation with the Icon-DMG pre-product; treatment at baseline of another caries lesion with an adhesive under rubber-dam isolation with the Prime Bont NT - Dentsply.
  Other Names: Infiltrant: Icon pre-product, DMG; Adhesive: Prime Bond NT, Dentsply
  Arms: Treatment with Infiltrant/Adhesive
Drug: Placebo — In this split-mouth design study, one of the three randomly selected approximal lesions will be treated with an infiltrant resin, one will be treated with an adhesive resin.
  Other Names: Placebo (cleaning of surface)
  Arms: Placebo, placebo treatment

SUMMARY:
The purpose of this study was to compare with a clinical randomized controlled split-mouth design study the changes in the therapeutic effect of infiltrating versus sealing proximal caries lesions and placebo treatment after 1, 2 and 3 years. The outcome was lesion progression, evaluated by radiographic techniques.

DETAILED DESCRIPTION:
Fissure sealing has been shown to inhibit not only the formation of occlusal caries but also to impede the progression of existing caries lesions. Lately, the concept of sealing caries to arrest lesion progression has been transferred to approximal surfaces. In a clinical study sealed approximal lesions showed significantly reduced progression after 18 month compared with those that were treated only with preventive measures.

The pores of enamel caries lesions provide diffusion pathways for acids and dissolved minerals. The aim of caries infiltration is to occlude these pores by infiltration with light curing resins in order to block the diffusion of acids into the lesion body. In contrast to caries sealing, caries infiltration aims to occlude the pores within the lesion rather then placing a diffusion barrier on the lesion surface. Several studies showed significantly reduced progression of infiltrated enamel lesions in demineralizing environments.

This split-mouth placebo-controlled randomized clinical trial was conducted on 16-35 year-old subjects in Bogotá, Colombia (IRB UB.162-2008).

The sample size calculated was of minimum 29 patients with 3 approximal lesions around the EDJ or in the dentin outer third.

The study population was students and patients from Unversidad El Bosque. Two visits were planned for the patients within same week. In the first visit baseline standardized bitewing radiographs were obtained and 3 proximal selected lesions were randomly selected. A clinical examination was conducted to assess DMF-T/S, and individual caries risk. Elastic orthodontic bands were placed between teeth of selected surfaces for elective temporary separation.

In the second visit selected lesions were visually classified with ICDAS criteria and activity status of lesions was assessed. The 3 lesions were randomly allocated to: A. Infiltration, B. Sealing, C. Placebo, and lesions were treated.

Subjects were clinically examined after one, two, and three years by two examiners (AC, JSL) blinded to the selected treatment groups and referral for operative treatment were done if needed. Standardized bitewing radiographs were made each year.

Lesions progression was assessed on radiographs by pair-wise reading by an external examiner blinded to groups. Additionally, after one year reading of images was conducted by digital-subtraction radiography of scanned images. For reproducibility assessment the examiner repeated 20% of radiograph readings by both methods one week after the first reading.

Statistical analysis Intra-examiner reliability for radiographs readings was assessed by unweighted kappa scores; caries experience (DMF-T/S), individual caries risk levels, ICDAS criteria, radiographic scores, and progression' status of selected lesions were reported descriptively.

The outcome variable of changes in lesion progression after 1, 2 and 3 years was assessed by pair-wise radiographic reading and after one year also by digital-subtraction radiography.

Differences in lesion progression between treatments at each follow-up were tested by the Cochran Q test and in case of significant difference between groups, by the McNemar Change test, including the therapeutic effect and the 95% confidence intervals [Siegel & Castellan, 1988].

In all tests p-values less than 0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were to have at least three caries proximal lesions on their posterior permanent teeth with a radiographic severity classification of the lesion score of 3 -Around the enamel dentin junction (EDJ) or 4 -Dentin-outer 1/3.

Exclusion Criteria:

* Under orthodontic treatment at enrollment
* Moving from the city (Bogota) in the following three years after commencing the study.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pair-wise radiographic lesion progression | 1, 2, and 3 years
  Changes in the therapeutic effect of infiltrating versus sealing proximal caries lesions and placebo treatment after 1, 2 and 3 years. The outcome was lesion progression, evaluated by radiographic techniques.

SECONDARY OUTCOMES:
Digital-subtraction radiography lesion progression | 1 year
  Changes in the therapeutic effect of infiltrating versus sealing proximal caries lesions and placebo treatment after 1 year. The outcome was lesion progression, evaluated by subtraction radiography.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Martignon, PhD, Study Chair — Universidad El Bosque, Bogotá, COlombia
Locations (1):
- Universidad El Bosque, Bogotá, D.c:, Colombia

REFERENCES:
- [Background] Martignon S, Ekstrand KR, Ellwood R. Efficacy of sealing proximal early active lesions: an 18-month clinical study evaluated by conventional and subtraction radiography. Caries Res. 2006;40(5):382-8. doi: 10.1159/000094282. PMID 16946605
- [Background] Martignon S, Tellez M, Santamaria RM, Gomez J, Ekstrand KR. Sealing distal proximal caries lesions in first primary molars: efficacy after 2.5 years. Caries Res. 2010;44(6):562-70. doi: 10.1159/000321986. Epub 2010 Nov 19. PMID 21088401
- [Background] Ekstrand KR, Bakhshandeh A, Martignon S. Treatment of proximal superficial caries lesions on primary molar teeth with resin infiltration and fluoride varnish versus fluoride varnish only: efficacy after 1 year. Caries Res. 2010;44(1):41-6. doi: 10.1159/000275573. Epub 2010 Jan 15. PMID 20090327
- [Derived] Martignon S, Ekstrand KR, Gomez J, Lara JS, Cortes A. Infiltrating/sealing proximal caries lesions: a 3-year randomized clinical trial. J Dent Res. 2012 Mar;91(3):288-92. doi: 10.1177/0022034511435328. Epub 2012 Jan 17. PMID 22257664